CLINICAL TRIAL: NCT00759343
Title: Stone Centre Urine and Serum Bank
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Other Study IDs: H06-00151
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Kidney Stones
Keywords: Kidney stones; urinary stone disease; urinary stones; urine; serum
MeSH Terms: conditions — Kidney Calculi; Urinary Calculi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Urine and serum of stone-forming individuals and non-stone forming controls will be banked for analysis of protein biomarkers and predisposing factors. Ureteral stents removed from patients that would otherwise be discarded will be processed and stored to assess for bacterial and biofilm adherence.
  Serum and Urine specimens will be collected, de-identified, and banked/retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: The control subjects of this study will be asked to undergo renal ultrasound examination, if available, or will be asked to complete a disease history form to determine the presence or lack of a kidney stone. Urine and serum will then be taken for storage until further analysis.
  Controls will be asked to undergo a screening renal ultrasound to ensure they are stone free, this will take approximately 45 minutes. If the controls are asked to complete the history form, this will not take more than 20 minutes. They will also give a blood and urine sample during this time to bring the total extra time up to at most 60 minutes for controls."
- Stone Group: The stone group will undergo standard diagnostic procedures for their condition and recovery process. Serum and urine for storage and analysis will be taken prior to stone treatment and 6 weeks following stone treatment. This will allow for the determination of differences in a stone patient's protein profile while they have their stone and after they are stone free. All patients will be required to have a stone patient metabolic evaluation which includes serum and urine testing. The analysis will focus on the serum and urine sample that they provide.
  The stone patient will be asked to undergo one extra tube of blood during their preoperative assessment which should only add a few seconds to their visit.

SUMMARY:
Purpose:

The purpose of the Stone Centre Serum and Urine Bank is to provide researchers with large numbers of serum and urine samples from kidney stone patients and controls for study of stone disease detection and treatment, and will take into account different genetic backgrounds, ages, and other patient factors to provide a broad sample size for the study of stone disease The Serum and Urine Bank will undoubtedly be an invaluable tool in the quest to understanding urinary stone disease.

Objective:

The objective of this research is to identify protein species or other compounds responsible for or contributing to kidney stone initiation and propagation.

DETAILED DESCRIPTION:
Background:

While great strides have been made in the surgical treatment of kidney stones, the means to identify high-risk patients for the prevention of kidney stones has lagged far behind. Urinary stone disease is a common problem, causes significant disability and sometimes death, and costs society 1.8 billion dollars each year. Therefore, it is important to identify those patients who are at risk or in the process of developing kidney stones and develop procedures which halt and/or prevent stone formation. Unfortunately, the current methods used for identifying such patients are inadequate. Kidney stone patients undergo urine and serum testing to attempt to identify substances that are either in excess or deficit in the body. The levels of these substances are then adjusted with diet modification and/or the use of medication. Often, patients who have corrected their abnormal values via diet or medications or others who have no identifiable risk factors continue to form stones. Clearly, current testing methods used to identify the continuous formation of stones are not enough, largely due to the fact that the causes of this disease are not completely understood.

There exists strong evidence supporting a role for proteins, both in promoting stone formation and in their prevention. Furthermore there may be hereditary factors (i.e. a family history) that may increase the risk of some patients becoming chronic kidney stone formers. This suggests a very complex cause of the disease and emphasizes the need and importance of identifying the genes and proteins involved in formation of stones.

Research Methods:

Urine and serum samples will be collected from study and control groups. Study group will be formed from confirmed kidney stone patients followed until post recovery, and the control group from healthy individuals. Control patients will have no history of kidney stone disease. Control subjects may be asked to undergo a screening renal ultrasound to ensure they are stone free.

If there is ureteral stent placed after surgery in stone patients, once it is removed, it is typically thrown into the garbage. With this study, it will be removed and the surface of the stent will be examined for crystals and adherent proteins. The collected samples will be submitted for SELDI analysis and to measure non-protein components. Each patient's serum sample will also be submitted for protein analysis. Other samples will be stored indefinitely until used. The urine, serum, and ureteral stents obtained in this study will be banked at -80C in a locked, secure area.

Recruitment:

Recruitment of study group will be through the Urology and Stone Clinic in the Diamond Health Care Centre at Vancouver General Hospital and Dr Joel Teichman's Practice at St Paul's Hospitals. Patients will be asked to participate by a urologist (Drs Chew, Teichman, Nigro, Fenster or Paterson) or the research coordinator. Control patients will be matched for age and sex to the study group. They will have no history of stone disease. The consent form will be provided to the participants by one of the investigators or a clinical research coordinator involved in the study. This will occur in one of the urology clinics.

Risks:

The risks involved are minimal; drawing blood can result in possible bleeding, fainting, bruising and infection. Urine collection has minimal risks.

Benefits:

There will not be any direct benefit from taking part in this urine and serum banking. We anticipate that the information gained will benefit others in the future and provide detection and treatment of urinary stone disease. No reimbursements or payments are being offered, as there will be no expenses to the patients as a result of the banking of urine and serum.

Confidentiality:

All samples will be coded to preserve anonymity of the subjects. Once distributed, the samples will be labeled only with the code. At no point in time will the patient identifiers leave the Stone Centre Serum and Urine Bank.

ELIGIBILITY:
Inclusion Criteria:

* Controls: age > 19 and no history of kidney stone disease);
* Study (Stone Patient): Age > 19, radiological evidence indicating presence of a current renal or ureteric stone.

Exclusion Criteria:

* Pregnancy,
* Positive Urine Culture,
* Active cancer,
* Recurrent urinary infections,
* Gross hematuria,
* Inability to provide informed consent,
* Investigator's refusal to include,
* CONTROLS ONLY:

  * Family history of stones,
  * History of stones

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Accepts patients with stone disease and healthy volunteers as controls
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-06; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
genetic factors in stone disease | one time sample
  We are to determine the genetic factors that contributes to kidney stone disease from the microbiome analysis of urine and serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Ben H. Chew, MD, FRCSC, Principal Investigator — University of British Columbia; Ryan Paterson, MD, Study Director — University of British Columbia; Howard Fenster, MD, Study Director — University of British Columbia; Caitlin Dobie, Study Director — University of British Columbia; Dirk Lange, MD, Study Director — University of British Columbia; Mark Nigro, MD, Study Director — University of British Columbia
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - UBC Hospital, Vancouver, British Columbia

REFERENCES:
- See also: Related Info — http://clinicaltrials.gov/ct2/show/NCT00199459